CLINICAL TRIAL: NCT01242514
Title: (OSKIRA-X): A Long-term Extension Study to Assess the Safety and Efficacy of Fostamatinib Disodium in the Treatment of Rheumatoid Arthritis
Brief Title: Evaluation of Long-term Safety and Effectiveness of Fostamatinib in the Treatment of Rheumatoid Arthritis (RA)
Acronym: OSKIRA-X
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: AZ decision to discontinue fostamatinib development in RA; rights to fostamatinib returned to Rigel Pharmaceuticals.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D4300C00005; 2010-020892-22 (EudraCT Number)
Record Dates: First submitted 2010-11-10; First posted 2010-11-17 (Estimated); Results first posted 2014-04-04 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2014-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; OSKIRA; Fostamatinib
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — fostamatinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): Oral treatment
  Interventions: Drug: Fostamatinib
- B (Experimental): Oral treatment
  Interventions: Drug: Fostamatinib
- C (Experimental): Oral treatment
  Interventions: Drug: Fostamatinib

INTERVENTIONS:
Drug: Fostamatinib — Fostamatinib 100mg twice daily
  Arms: A
Drug: Fostamatinib — Fostamatinib 150mg once daily
  Arms: B
Drug: Fostamatinib — Fostamatinib 100mg once daily
  Arms: C

SUMMARY:
The purpose of this study is to evaluate the long term safety and tolerability of fostamatinib in patients with rheumatoid arthritis (RA).

ELIGIBILITY:
Inclusion Criteria:

* Patients who have successfully completed a qualifying study (D4300C00001, D4300C00002, D4300C00003 or D4300C00004) with fostamatinib
* Patients who have participated in a qualifying study and who have been classified as non-responders due to pre-defined lack of efficacy at Week 12 (D4300C00001, D4300C00002, D4300C00003).

Exclusion Criteria:

* Premature withdrawal from the qualifying study (D4300C00001, D4300C00002, D4300C00003 and D4300C00004)
* Females who are pregnant or breast feeding
* Poorly controlled hypertension
* Significant liver function test abnormalities or physical symptoms of hepatotoxicity
* Significant infection
* Gastrointestinal intolerance
* Cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1917 (Actual)
Dates: Start 2011-01; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Chris O'Brien, MD PhD, Study Director — AstraZeneca
Locations (308):
- United States (116):
  - Research Site, Anniston, Alabama
  - Research Site, Birmingham, Alabama
  - Research Site, Huntsville, Alabama
  - Research Site, Tuscaloosa, Alabama
  - Research Site, Glendale, Arizona
  - Research Site, Mesa, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Scottsdale, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Hot Springs, Arkansas
  - Research Site, Anaheim, California
  - Research Site, Fountain Valley, California
  - Research Site, Huntington Beach, California
  - Research Site, La Jolla, California
  - Research Site, Long Beach, California
  - Research Site, Palo Alto, California
  - Research Site, Roseville, California
  - Research Site, Santa Maria, California
  - Research Site, Santa Monica, California
  - Research Site, Torrance, California
  - Research Site, Upland, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Bridgeport, Connecticut
  - Research Site, Danbury, Connecticut
  - Research Site, Trumbull, Connecticut
  - Research Site, Lewes, Delaware
  - Research Site, Boca Raton, Florida
  - Research Site, Brandon, Florida
  - Research Site, Daytona Beach, Florida
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Ocala, Florida
  - Research Site, Orlando, Florida
  - Research Site, Palm Harbor, Florida
  - Research Site, Pinellas Park, Florida
  - Research Site, Tampa, Florida
  - Research Site, Tavares, Florida
  - Research Site, Venice, Florida
  - Research Site, Zephyrhills, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Canton, Georgia
  - Research Site, Decatur, Georgia
  - Research Site, Lawrenceville, Georgia
  - Research Site, Macon, Georgia
  - Research Site, Marietta, Georgia
  - Research Site, Idaho Falls, Idaho
  - Research Site, Chicago, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, South Bend, Indiana
  - Research Site, Cedar Rapids, Iowa
  - Research Site, Bowling Green, Kentucky
  - Research Site, Elizabethtown, Kentucky
  - Research Site, Cumberland, Maryland
  - Research Site, Frederick, Maryland
  - Research Site, Hagerstown, Maryland
  - Research Site, Oxon Hill, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Fall River, Massachusetts
  - Research Site, Worcester, Massachusetts
  - Research Site, Kalamazoo, Michigan
  - Research Site, Lansing, Michigan
  - Research Site, Saint Clair Shores, Michigan
  - Research Site, Eagan, Minnesota
  - Research Site, Flowood, Mississippi
  - Research Site, Florissant, Missouri
  - Research Site, Richmond Heights, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Kalispell, Montana
  - Research Site, Omaha, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Freehold, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Las Cruces, New Mexico
  - Research Site, Albany, New York
  - Research Site, Brooklyn, New York
  - Research Site, Cooperstown, New York
  - Research Site, Olean, New York
  - Research Site, Roslyn, New York
  - Research Site, Smithtown, New York
  - Research Site, Syracuse, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Research Triangle Park, North Carolina
  - Research Site, Dayton, Ohio
  - Research Site, Mayfield Village, Ohio
  - Research Site, Perrysburg, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Lake Oswego, Oregon
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Erie, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Waxford, Pennsylvania
  - Research Site, West Reading, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Orangeburg, South Carolina
  - Research Site, Rapid City, South Dakota
  - Research Site, Hixson, Tennessee
  - Research Site, Jackson, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Amarillo, Texas
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Katy, Texas
  - Research Site, Lubbock, Texas
  - Research Site, Mesquite, Texas
  - Research Site, Nassau Bay, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Chesapeake, Virginia
  - Research Site, Tacoma, Washington
- Argentina (10):
  - Research Site, Buenos Aires, Buenos Aires F.D.
  - Research Site, Ciudad Autonoma Bs As, CBA
  - Research Site, Córdoba, CRD
  - Research Site, San Juan, San Juan Province
  - Research Site, Rosario, Santa Fe Province
  - Research Site, San Miguel de Tucumán, TUC
  - Research Site, Caba Buenos Aires
  - Research Site, Ciudad Autonoma Bs As
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Quilmes
- Australia (3):
  - Research Site, Camperdown, New South Wales
  - Research Site, Southport, Queensland
  - Research Site, Cairns
- Belgium (5):
  - Research Site, Ghent, Belgium
  - Research Site, Liège, Belgium
  - Research Site, Brussels
  - Research Site, Gilly
  - Research Site, Yvoir
- Brazil (5):
  - Research Site, Goiânia, Goiás
  - Research Site, Curitiba, Paraná
  - Research Site, Recife, Pernambuco
  - Research Site, São Paulo, São Paulo
  - Research Site, Rio de Janeiro
- Bulgaria (4):
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Sevlievo
  - Research Site, Sofia
- Canada (15):
  - Research Site, Edmonton, Alberta
  - Research Site, Victoria, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Bowmanville, Ontario
  - Research Site, Etobicoke, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Pointe-Claire, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Rimouski, Quebec
  - Research Site, Trois-Rivières, Quebec
- Chile (2):
  - Research Site, Osorno, Los Lagos Region
  - Research Site, Santiago
- Colombia (3):
  - Research Site, Barranquilla, Atlántico
  - Research Site, Bogota, Cundinamarca
  - Research Site, Bucaramanga, Santander Department
- Czechia (14):
  - Research Site, Brno
  - Research Site, Bruntál
  - Research Site, Česká Lípa
  - Research Site, České Budějovice
  - Research Site, Hlučín
  - Research Site, Hostivice
  - Research Site, Kladno
  - Research Site, Liberec
  - Research Site, Ostrava
  - Research Site, Ostrava - Trebovice
  - Research Site, Prague
  - Research Site, Sokolov
  - Research Site, Terezín
  - Research Site, Zlín
- Estonia (3):
  - Research Site, Pärnu
  - Research Site, Tallinn
  - Research Site, Tartu
- Research Site, Orléans, France
- Germany (10):
  - Research Site, Aachen, North Rhine-Westphalia
  - Research Site, Halle, Saxony
  - Research Site, Cologne
  - Research Site, Erlangen
  - Research Site, Frankfurt
  - Research Site, Hamburg
  - Research Site, Heidelberg
  - Research Site, Herne
  - Research Site, Leipzig
  - Research Site, München
- Hungary (8):
  - Research Site, Balatonfüred
  - Research Site, Békéscsaba
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Makó
  - Research Site, Sopron
  - Research Site, Szentes
  - Research Site, Zalaegerszeg-pozva
- India (14):
  - Research Site, Hyderabad, Andhra Pradesh
  - Research Site, Secunderabad, Andhra Pradesh
  - Research Site, Ahmedabad, Gujarat
  - Research Site, Gandhinagar, Gujarat
  - Research Site, Vadodara, Gujarat
  - Research Site, Bangalore, Karnataka
  - Research Site, Mangalore, Karnataka
  - Research Site, Udupi, Karnataka
  - Research Site, Mumbai, Maharashtra
  - Research Site, Pune, Maharashtra
  - Research Site, Nagpur, Maharshtra
  - Research Site, Coimbatore, Tamil Nadu
  - Research Site, Madurai, Tamil Nadu
  - Research Site, Lucknow, Uttar Pradesh
- Israel (5):
  - Research Site, Ashkelon
  - Research Site, Haifa
  - Research Site, Kfar Saba
  - Research Site, Ramat Gan
  - Research Site, Rehovot
- Italy (3):
  - Research Site, Iesi, AN
  - Research Site, Udine, UD
  - Research Site, Varese, VA
- Latvia (3):
  - Research Site, Liepāja
  - Research Site, Riga
  - Research Site, Valmiera
- Lithuania (3):
  - Research Site, Kaunas
  - Research Site, Klaipėda
  - Research Site, Šiauliai
- Mexico (8):
  - Research Site, Chihuahua City, Chihuahua
  - Research Site, Saltillo, Coahuila
  - Research Site, Mexicali, Estado de Baja California
  - Research Site, Guadalajara, Jalisco
  - Research Site, Mexico City, Mexico City
  - Research Site, San Luis Potosi, Mexico
  - Research Site, Monterrey, Nuevo León
  - Research Site, Obrergon, Sonora
- Peru (5):
  - Research Site, Arequipa, Arequipa
  - Research Site, Lima, Lima Province
  - Research Site, Pueblo Libre, Lima region
  - Research Site, San Borja, Lima region
  - Research Site, San Isidro, Lima region
- Poland (10):
  - Research Site, Bytom
  - Research Site, Chełm Śląski
  - Research Site, Grodzisk Mazowiecki
  - Research Site, Kalisz
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Warsaw
  - Research Site, Wroclaw
  - Research Site, Żyrardów
- Portugal (4):
  - Research Site, Aveiro
  - Research Site, Coimbra
  - Research Site, Lisbon
  - Research Site, Porto
- Romania (2):
  - Research Site, Ploieşti, Prahova
  - Research Site, Brăila
- Russia (7):
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Petrozavodsk
  - Research Site, Ryazan
  - Research Site, Saint Petersburg
  - Research Site, Voronezh
  - Research Site, Yaroslavl
- Serbia (4):
  - Research Site, Belgrade
  - Research Site, Kragujevac
  - Research Site, Niška Banja
  - Research Site, Novi Sad
- Slovakia (6):
  - Research Site, Bratislava, Slovakia
  - Research Site, Žilina, Slovakia
  - Research Site, Poprad
  - Research Site, Rimavská Sobota
  - Research Site, Ružomberok
  - Research Site, Trnava
- South Africa (7):
  - Research Site, Panorama, Cape Town
  - Research Site, Port Elizabeth, E Cape
  - Research Site, Kempron Park, Gauteng
  - Research Site, Pretoria, Gauteng
  - Research Site, Durban, KwaZulu-Natal
  - Research Site, Cape Town, Western Cape
  - Research Site, Stellenbosch
- Spain (2):
  - Research Site, Mérida, Extremadura
  - Research Site, Barcelona
- Ukraine (12):
  - Research Site, Donetsk
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv
  - Research Site, Kyiv
  - Research Site, Luhansk
  - Research Site, Lutsk
  - Research Site, Lviv
  - Research Site, Odesa
  - Research Site, Simferopol
  - Research Site, Vinnytsia
  - Research Site, Zaporizhzhya
  - Research Site, Zaporyzhzhya
- United Kingdom (14):
  - Research Site, Bracknell, Berkshire
  - Research Site, Warrington, Cheshire
  - Research Site, London, Greater London
  - Research Site, Maidstone, Kent
  - Research Site, Eastbourne, Sussex
  - Research Site, Solihull, West Midlands
  - Research Site, Basingstoke
  - Research Site, Cambridge
  - Research Site, Christchurch
  - Research Site, Ipswich
  - Research Site, Metropolitan Borough of Wirral
  - Research Site, Nottingham
  - Research Site, Stoke-on-Trent
  - Research Site, Westcliff-on-the Sea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total of 1917 enrolled patients: 1346, 357 & 214 were allocated to the 100 mg twice daily (bid), 150 mg once daily (qd) and 100 mg qd groups, respectively (1343, 357 & 212 received at least 1 dose of investigational product). As this was a long-term extension study no specific end date was given. As such no patients were recorded as completers.
Pre-assignment Details: A total of 5 patients did not receive treatment.
Groups:
- Fostamatinib 100 mg Bid; Fostamatinib 150 mg qd; Fostamatinib 100 mg qd: Oral treatment
Period: Overall Study
Arm/Group | Fostamatinib 100 mg Bid | Fostamatinib 150 mg qd | Fostamatinib 100 mg qd
Started | 1343 (Patients who received treatment) | 357 (Patients who received treatment) | 212 (Patients who received treatment)
Enrolled But Did Not Receive Treatment | 3 (Other) | 0 | 2 (Adverse event/other)
Completed | 0 (Due to project closure.) | 0 (Due to project closure.) | 0 (Due to project closure.)
Not Completed | 1343 | 357 | 212
Not completed — e.g., project closure | 1042 | 305 | 171
Not completed — Subject decision | 33 | 8 | 2
Not completed — Severe non-compliance to protocol | 5 | 2 | 1
Not completed — Lack of therapeutic response | 99 | 16 | 10
Not completed — Dev. of study specific discont. criteria | 21 | 3 | 5
Not completed — Lost to Follow-up | 14 | 5 | 4
Not completed — Adverse Event | 129 | 18 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fostamatinib 100 mg Bid | Fostamatinib 150 mg qd | Fostamatinib 100 mg qd | Total
Number analyzed (Participants) | 1343 | 357 | 212 | 1912
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (12.0) | 53 (11.6) | 53 (11.3) | 53 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1086 | 297 | 193 | 1576
  Male | 257 | 60 | 19 | 336
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 1092 | 278 | 141 | 1511
  Black or African American | 63 | 11 | 6 | 80
  Asian | 40 | 12 | 7 | 59
  American Indian or Alaska Native | 20 | 11 | 6 | 37
  Indian or Pakistani | 54 | 15 | 22 | 91
  Other | 74 | 30 | 30 | 134

OUTCOME MEASURES:

1. Secondary Outcome: Mean DAS28-CRP Score
Description: DAS28-CRP: Disease Activity Score based on a count of swollen and tender joints (out of 28 joints), blood test measures of inflammation (CRP) and the patient's own assessment. Scores can take any positive value with a lower value indicating a better clinical condition. Number of participants are those with data at entry to this study (Week 0). As no imputation was applied, the numbers at subsequent visits are lower. bid = twice daily, CRP = C-reactive protein, qd = once daily
Time Frame: Weeks 0, 12, 24, 36 and 52
Population: The full analysis set includes those patients who received at least 1 dose of investigational product, and were summarised according to treatment first received in this study (intention-to-treat principle).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Fostamatinib 100 mg Bid | Fostamatinib 150 mg qd | Fostamatinib 100 mg qd
Number analyzed (Participants) | 1247 | 336 | 198
Units on a scale
  Week 0 (n=1247, 336, 198) | 4.5 (1.58) [0.23 to 0.90] | 3.8 (1.24) [0.14 to 0.84] | 3.9 (1.27) [-0.12 to 0.56]
  Week 12 (n=1018, 288, 160) | 3.8 (1.34) | 3.6 (1.19) | 3.7 (1.21)
  Week 24 (n=800, 230 126) | 3.8 (1.30) | 3.7 (1.24) | 3.6 (1.19)
  Week 36 (n=581, 148, 68) | 3.9 (1.32) | 3.7 (1.24) | 3.9 (1.07)
  Week 52 (n=290, 28, 14) | 4.0 (1.25) | 3.8 (1.37) | 3.6 (1.22)

2. Primary Outcome: Percentage of Patients Who Had at Least 1 Adverse Event in Any Category
Description: AE = adverse event, bid = twice daily, IP = investigational product, qd = once daily, SAE = serious adverse event
Time Frame: Entry in extension to end of study (variable duration; maximum 109 weeks)
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Fostamatinib 100 mg Bid | Fostamatinib 150 mg qd | Fostamatinib 100 mg qd
Number analyzed (Participants) | 1343 | 357 | 212
Percentage of patients
  Any AE | 74.4 | 70.3 | 69.8
  Any AE with outcome of death | 0.7 | 0.3 | 0.5
  Any SAE (including events with outcome of death) | 11.4 | 8.7 | 5.7
  Any AE leading to discontinuation of IP | 10.5 | 5.9 | 9.9

3. Secondary Outcome: Mean mTSS Score
Description: mTSS: modified total sharp score, a measure of structural progression based upon X-rays. Hand and foot joints are scored for erosions and joint space narrowing and the results summed to give a value between 0 and 488. A higher value represents more serious progression of the disease. Number of participants are those with data at entry to this study (Week 0). As no imputation was applied, the numbers at subsequent visits are lower. bid = twice daily, N/A = not applicable, qd = once daily
Time Frame: Weeks 0 and 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Fostamatinib 100 mg Bid | Fostamatinib 150 mg qd | Fostamatinib 100 mg qd
Number analyzed (Participants) | 480 | 73 | 37
Units on a scale
  Week 0 (n=480, 73, 37) | 30.5 (47.73) | 22.2 (32.89) | 20.8 (46.60)
  Week 52 (n=223, 1, 6) | 30.1 (46.83) | 0.5 (NA) — Measures of spread are not defined for treatment groups containing a single patient. | 37.3 (67.70)

4. Secondary Outcome: Mean HAQ-DI Score
Description: HAQ-DI: Health Assessment Questionnaire - Disability Index, a measure of physical function. The HAQ-DI score is then calculated by summing the category scores from 8 sub-categories (ie, scores for patient ability in dressing and grooming, rising, eating, walking, hygiene, reach, grip and common daily activities) and dividing by the number of categories completed. The HAQ-DI score takes values between 0 and 3, with a higher score indicating greater disability. Number of participants are those with data at entry to this study (Week 0). As no imputation was applied, the numbers at subsequent visits are lower. bid = twice daily, qd = once daily
Time Frame: Weeks 0, 12, 24, 36 and 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Fostamatinib 100 mg Bid | Fostamatinib 150 mg qd | Fostamatinib 100 mg qd
Number analyzed (Participants) | 1271 | 342 | 201
Units on a scale
  Week 0 (n=1271, 342, 201) | 1.2 (0.69) | 1.0 (0.64) | 1.0 (0.62)
  Week 12 (n=1061, 298, 166) | 1.1 (0.68) | 1.0 (0.63) | 1.0 (0.63)
  Week 24 (n=817, 238, 132) | 1.1 (0.68) | 1.0 (0.67) | 0.9 (0.55)
  Week 36 (n=587, 149, 71) | 1.1 (0.67) | 1.0 (0.65) | 1.1 (0.62)
  Week 52 (n=296, 28, 14) | 1.2 (0.68) | 1.1 (0.64) | 1.0 (0.73)

ADVERSE EVENTS:
Arm/Group | FOSTA 100 MG BID | FOSTA 100 MG QD | FOSTA 150 MG QD
Serious Adverse Events (participants affected / at risk) | 153/1343 | 12/212 | 31/357
Other Adverse Events (participants affected / at risk) | 466/1343 | 68/212 | 98/357
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOSTA 100 MG BID (N=1343) | FOSTA 100 MG QD (N=212) | FOSTA 150 MG QD (N=357)
SPLENIC INFARCTION (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
ANGINA UNSTABLE (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
BRADYCARDIA (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
CARDIAC FAILURE CHRONIC (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
CARDIOMYOPATHY (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
GOITRE (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
RETINAL DETACHMENT (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
ACUTE ABDOMEN (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
BARRETT'S OESOPHAGUS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
COLITIS (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
COLITIS MICROSCOPIC (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
COLONIC STENOSIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
GASTRIC ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
GASTRITIS EROSIVE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
HAEMATEMESIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
ILEITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
ILEUS (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
INGUINAL HERNIA (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
OESOPHAGEAL ACHALASIA (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
PANCREATIC PSEUDOCYST (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
DEVICE DISLOCATION (General disorders) | 1 (1) | 0 (0) | 0 (0)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1 (1) | 0 (0) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 3 (3) | 1 (1) | 0 (0)
BILE DUCT OBSTRUCTION (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
BILIARY COLIC (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
CHOLECYSTITIS (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
CHOLECYSTITIS CHRONIC (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
CHOLELITHIASIS (Hepatobiliary disorders) | 4 (4) | 0 (0) | 0 (0)
GALLBLADDER POLYP (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
POST CHOLECYSTECTOMY SYNDROME (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
ANAPHYLACTIC SHOCK (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
FOOD ALLERGY (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
HYPERSENSITIVITY (Immune system disorders) | 2 (2) | 0 (0) | 0 (0)
ABSCESS LIMB (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
APPENDICITIS (Infections and infestations) | 4 (4) | 0 (0) | 0 (0)
ARTHRITIS BACTERIAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
BACTERIAL PYELONEPHRITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
BACTERIAL SEPSIS (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
BRONCHOPNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
CELLULITIS (Infections and infestations) | 6 (7) | 1 (1) | 0 (0)
CYTOMEGALOVIRUS INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
ENTEROCOLITIS BACTERIAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
ENTEROCOLITIS VIRAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
ERYSIPELAS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
GANGRENE (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
GASTROENTERITIS BACTERIAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
GASTROENTERITIS VIRAL (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
HERPES ZOSTER (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
INTERVERTEBRAL DISCITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
LIVER ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
LUNG ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OSTEOMYELITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTITIS EXTERNA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PANCREATITIS VIRAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PERITONITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 5 (5) | 1 (1) | 1 (1)
PNEUMONIA BACTERIAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA VIRAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PULMONARY TUBERCULOSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
SUBCUTANEOUS ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
URINARY TRACT INFECTION BACTERIAL (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
UROSEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
WOUND INFECTION BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
WOUND SEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1)
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
JOINT INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
PATELLA FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
TENDON RUPTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
ULNA FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
WRIST FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
LIVER FUNCTION TEST ABNORMAL (Investigations) | 1 (1) | 0 (0) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
HIP DEFORMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
INTERVERTEBRAL DISC DISORDER (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
INTERVERTEBRAL DISC DISPLACEMENT (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 0 (0)
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
OSTEITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 6 (8) | 0 (0) | 2 (2)
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 9 (11) | 0 (0) | 0 (0)
SJOGREN'S SYNDROME (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
SPONDYLOLISTHESIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
SYNOVITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
BENIGN NEOPLASM OF PROSTATE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
BENIGN SOFT TISSUE NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
CERVIX CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
COLORECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
LIPOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
LUNG SQUAMOUS CELL CARCINOMA STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
PANCREATIC NEUROENDOCRINE TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
RENAL CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 1 (1)
VAGINAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
APHASIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
CAROTID ARTERY STENOSIS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
CONVULSION (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
DYSARTHRIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
HAEMORRHAGIC STROKE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
HYPERTENSIVE ENCEPHALOPATHY (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
HYPOGLYCAEMIC COMA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
ISCHAEMIC STROKE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
LUMBAR RADICULOPATHY (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
POSTERIOR REVERSIBLE ENCEPHALOPATHY SYNDROME (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
RADICULITIS LUMBOSACRAL (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
SCIATICA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 3 (3) | 0 (0) | 2 (2)
TENSION HEADACHE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
VITH NERVE PARALYSIS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
ADJUSTMENT DISORDER (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
ALCOHOL ABUSE (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
DEPRESSION (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
CALCULUS URETERIC (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
CALCULUS URINARY (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0)
RENAL IMPAIRMENT (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
URINARY BLADDER POLYP (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
ADENOMYOSIS (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
OVARIAN CYST (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
UTERINE POLYP (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
HYPERVENTILATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
DIGITAL ULCER (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
ERYTHEMA MULTIFORME (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
TOXIC EPIDERMAL NECROLYSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
AORTIC ANEURYSM RUPTURE (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
AORTIC STENOSIS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
AORTIC THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
ARTERIAL THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
FEMORAL ARTERY OCCLUSION (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
PERIPHERAL ISCHAEMIA (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
THROMBOPHLEBITIS SUPERFICIAL (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOSTA 100 MG BID (N=1343) | FOSTA 100 MG QD (N=212) | FOSTA 150 MG QD (N=357)
DIARRHOEA (Gastrointestinal disorders) | 202 (268) | 28 (40) | 43 (61)
NASOPHARYNGITIS (Infections and infestations) | 86 (102) | 15 (16) | 28 (31)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 116 (155) | 19 (22) | 30 (35)
HYPERTENSION (Vascular disorders) | 166 (197) | 14 (15) | 20 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on the PI is that the sponsor can review and comment on results communications prior to publication. Sponsor will be allowed a review period of at least 60 days from submission but can request that publication be delayed for a period up to 6 months. Any reasonable comments made by the sponsor will be incorporated by the PI into the publication.